CLINICAL TRIAL: NCT04615936
Title: Methylene Blue-mediated Photodisinfection for SARS-CoV-2 in the Upper Respiratory Tract
Brief Title: Nasal Photodisinfection COVID-19 Proof of Concept Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NasalPDF001
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; Corona Virus Infection; SARS-CoV 2
Keywords: COVID-19; SARS-CoV-2; coronavirus; influenza; photodisinfection; nasal photodisinfection
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Influenza, Human

STUDY DESIGN:
Intervention Model Description: There is only a single group of patients in the study who will undergo treatment. There is a small sub group/'nil' group of 3 healthcare workers that will not be undergoing the treatment but will instead be doing multiple nasal swabbing in the course of 5 days.
Masking Description: N/A- masking not required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methylene Blue-Photodisinfection (Experimental): The Health-Canada approved Steriwave system (Ondine Biomedical, BC) will be used to deliver the Methylene Blue-Photodisinfection (MB-PDF) to the anterior nares.
  Interventions: Other: Methylene-Blue Photodisinfection

INTERVENTIONS:
Other: Methylene-Blue Photodisinfection — Participants will receive a pre-treatment nasal swab followed MB-PDF, this involves an MB nasal spray, followed by five minutes of red-light exposure into each nostril. Ten minutes after the treatment, a post treatment nasal swab will be performed.

SUMMARY:
The study proposes to test photodisinfection (PDF) on SARS-CoV-2 in the nose. The study will use Health Canada approved Steriwave™ Nasal Decolonization (ND) in he nostril of patients infected with SARS-CoV-2. Participants are swabbed for SARS-CoV-2 before and after the PDF treatment. For the study, a small group of healthcare workers who have tested positive for SARS-CoV-2 will be included. They will not undergo the treatment but will need to swab their noses multiple times over the next 5 days. This nil group will provide the effect (if any) of swabbing SARS-CoV-2 levels in the nose.

DETAILED DESCRIPTION:
The study proposes to test photodisinfetion (PDF) on levels of SARS-CoV-2 in the nose. The study will use Health Canada approved Steriwave™ Nasal Decolonization (ND) in patients infected with SARS-CoV-2 . Currrently, PDF is being used at some institutions before surgery to lower the risk of postoperative infection. PDF uses a Methylene Blue (MB) nasal spray, followed by 5 minutes of red-light exposure through a small light-diffusing applicator. This will need to be placed into each nostril. Participants are swabbed for SARS-CoV-2 before and after treatment. In addition to the patients testing positive for SARS-CoV-2, there will also be a small group of healthcare workers who have tested positive that will be included. Though they are not undergoing treatment, they will swab their own noses multiple times over a period of 5 days. This will allow us to evaluate the effect (if any) of swabbing on SARS-CoV-2 levels in the nose. The study hypothesis is that MB-mediated PDF will show the ability to kill SARS-CoV-2 which will consequently confirm its efficacy as a first line defense against the virus.

ELIGIBILITY:
Inclusion Criteria (patient population):

* Recent SARS-CoV-2+ diagnosis
* Present in hospital

Inclusion Criteria (healthcare workers):

* Recent SARS-CoV-2+ diagnosis
* Ability to self-administer nasal swabs

Exclusion Criteria (patient population):

* Immediate requirement for intubation (i.e. emergency airway) or inability to maintain independent oral airway

Exclusion Criteria (healthcare workers):

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
RT-qPCR | 30 minutes
  The main endpoint is microbiological; RT-qPCR will be conducted on the pre and post treatment swabs and the change in cycle threshold value will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Cari Whyne, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lobo CS, Rodrigues-Santos P, Pereira D, Nunez J, Trepa JCD, Sousa DL, Lourenco JV, Coelho MF, de Almeida LP, da Cunha JS, Arnaut LG. Photodynamic disinfection of SARS-CoV-2 clinical samples using a methylene blue formulation. Photochem Photobiol Sci. 2022 Jun;21(6):1101-1109. doi: 10.1007/s43630-022-00202-6. Epub 2022 Mar 19. PMID 35304729